CLINICAL TRIAL: NCT06649773
Title: A Study to Evaluate the Efficacy and Safety of Noiiglutide Injection in Type 2 Diabetes Patients Who Received Metformin in Combination With or Without Another Oral Hypoglycemic Drug for Poor Blood Glucose Control -- a Phase III Clinical Trial of Multicenter, Randomized, Double-blind, Placebo Parallel Control
Brief Title: The Experiment of Noiiglutide Injection in Type 2 Diabetes Patients
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR20004-302
Record Dates: First submitted 2024-10-08; First posted 2024-10-21 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Noiiglutide Injection (Experimental)
  Interventions: Drug: Noiiglutide Injection
- Noiiglutide Placebo (Placebo Comparator)
  Interventions: Drug: Noiiglutide Placebo

INTERVENTIONS:
Drug: Noiiglutide Injection — Experimental group
  Arms: Noiiglutide Injection
Drug: Noiiglutide Placebo — Placebo Comparator group
  Arms: Noiiglutide Placebo

SUMMARY:
This study aims to confirm that SHR20004 is more effective than placebo in controlling blood glucose in patients with type 2 diabetes. Evaluate the efficacy, safety, and pharmacokinetics of SHR20004 after 24 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria

1. Male or female, on the day of signing the informed consent form, aged between 18 and 75 years old;
2. During screening, according to the diagnostic criteria of the Chinese Guidelines for the Prevention and Treatment of Type 2 diabetes (2020 Edition), T2DM has a history of ≥ 3 months;
3. When screening, 7.5% ≤ HbA1c ≤ 10.0% (tested by local laboratory);
4. When filtering, 1) Metformin monotherapy for stable treatment for ≥ 3 months and daily dose ≥ 1500 mg or maximum tolerated dose (≥ 1000 mg); Or 2) Metformin combined with another domestically approved oral hypoglycemic drug for stable treatment for ≥ 3 months. Metformin is administered at the aforementioned dose, while the dose of the other oral hypoglycemic drug is ≥ half of the maximum approved dose or the maximum tolerated dose as indicated in the instructions. Another type of oral hypoglycemic drug must exclude drugs containing GLP-1 RA components (including multi-target drugs) and DPP-4 inhibitors;
5. When screening, 19.0 kg/m2 ≤ Body Mass Index (BMI) ≤ 45.0 kg/m2;
6. Capable and willing to comply with the protocol, including self-monitoring of blood glucose, recording participant diaries, and using pre filled injection pens;
7. From the signing of the informed consent form until 2 weeks after the last administration, the subject (including partner) has no plans to have children and is willing to use the high-efficiency contraceptive measures specified in the protocol.

Exclusion Criteria

1. The researchers suspect that the subjects may be allergic to the investigational drug;
2. Discontinuation of GLP-1 RA treatment due to safety/tolerability reasons or lack of effectiveness reasons in the past (excluding cases where GLP-1 RA is discontinued due to non efficacy or non safety reasons such as economic reasons, and no GLP-1 RA has been used within the past 3 months before screening);
3. Before screening, any of the following drugs or treatments were used:

   1. Have participated in any clinical trial of a drug within the first 3 months or 5 half lives (whichever is longer) before screening (has entered the randomization phase);
   2. Within 3 months, there has been drug or alcohol abuse that, according to the researcher's judgment, may affect the participation or status of the subjects in the trial, resulting in an impact on the use of trial drugs or compliance during the trial process;
   3. Screening for long-term (continuous 7 days or more) intravenous or oral administration of corticosteroids received within the previous 3 months;
   4. Within the first 3 months of screening, individuals who have used drugs with weight control effects, undergone surgeries that can cause weight instability, or experienced significant changes in weight (with a difference of ≥ 5 kg between maximum and minimum weight), or are currently on a weight loss plan and not in the maintenance phase;
   5. According to the researchers' judgment, any drug that may interfere with the interpretation of efficacy and safety data, or any drug known to have common toxic reactions to major organs, has been used within the previous month before screening;
4. History or evidence of any of the following diseases before screening:

   1. Type 1 diabetes, diabetes with single gene mutation, diabetes caused by pancreatic injury or other secondary diabetes, such as diabetes caused by Cushing's syndrome or acromegaly;
   2. There are high-risk factors that may lead to pancreatitis, such as a history of acute or chronic pancreatitis, a history of symptomatic gallbladder disease (excluding post cholecystectomy), and a history of pancreatic injury;
   3. A personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia type 2;
   4. There is a clinically relevant history of gastrointestinal disorders, accompanied by persistent nausea and vomiting, including but not limited to: gastroesophageal reflux disease with gastroparesis within the 6 months prior to screening, requiring treatment, unstable (worsening) or poorly controlled (persistent nausea and vomiting); Surgical history that may affect gastric emptying;
   5. Screening for severe hypoglycemic events or recurrent hypoglycemic events within the previous 6 months (≥ 3 hypoglycemic events within a week, or other hypoglycemic events determined by the researcher);
   6. Having obvious hematological disorders (such as aplastic anemia, myelodysplastic syndrome) or any disease that causes hemolysis or red blood cell instability (such as malaria);
   7. There are serious chronic complications of diabetes or there is a risk of acute complications within 6 months, and the investigator believes that it is not suitable to participate in this trial;
   8. Any organ system malignant tumor that has been treated or not treated within 5 years, regardless of evidence of local recurrence or metastasis, except for local basal cell carcinoma of the skin;
   9. Suffering from cardiovascular disease, defined as: having congestive heart failure (NYHA III-IV), unstable angina, stroke, myocardial infarction, or coronary revascularization within the first 6 months of screening; Plan to undergo coronary artery, carotid artery, or peripheral artery revascularization during screening;
   10. Systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg;
   11. There is a history of thyroid disease that cannot be controlled with stable drug dosage, and it has been determined by the researchers to affect the safety or efficacy of the subjects;
   12. Serious trauma or infection that may affect blood sugar control has occurred within one month;
5. During screening, laboratory tests showed the following situations:

   1. Fasting venous glucose ≥ 13.9 mmol/L;
   2. Serum amylase and/or serum lipase>3 times the upper limit of normal (ULN);
   3. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST)>3 × ULN;
   4. Moderate (3b) or severe renal failure or renal insufficiency (estimated glomerular filtration rate [eGFR] calculated using the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula<45 mL/min/1.73 m2) or in compliance with contraindications for metformin;
   5. Urinary albumin/creatinine ratio (UACR) ≥ 300 mg/g;
   6. Total bilirubin>2.0 × ULN;
   7. Calcitonin ≥ 50 ng/L;
   8. Triglycerides ≥ 5.7 mmol/L.
6. Abnormal 12 lead electrocardiograms with clinical significance during screening, such as grade II or III atrioventricular block (excluding right bundle branch block), long QT syndrome or QTc>500 ms, severe arrhythmia, etc. (mild T wave and ST segment changes may not be ruled out if the researcher judges that the subject's clinical symptoms are not obvious) in the absence of a pacemaker;
7. Within the first 4 weeks of screening, the amount of blood donated or lost is ≥ 400 mL, or a blood transfusion has been received;
8. Pregnant or lactating women, as well as fertile men or women who are unwilling to use contraception during the study period;
9. The researchers believe that the subjects have any other factors that may affect the efficacy or safety evaluation of this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2024-10-25 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes in glycated hemoglobin (HbA1c) relative to baseline at week 24 in SHR20004 compared to placebo. | Week 26

SECONDARY OUTCOMES:
The proportion of subjects who achieve the HbA1c target value (<7.0%) | Week 26
The proportion of subjects who achieve the HbA1c target value (≤ 6.5%) | Week 26
Changes in fasting plasma glucose relative to baseline | Week 26
Changes in fasting body weight relative to baseline | Week 26
Changes in plasma glucose levels relative to baseline 2 hours after meals | Week 26
7-point self-test of blood glucose (SMBG) spectrum relative to baseline changes | Week 26
Changes in blood pressure relative to baseline | Week 26
Changes in fasting insulin relative to baseline | Week 26
Changes in C-peptide relative to baseline | Week 26
Changes in insulin levels relative to baseline 2 hours after meals | Week 26
Changes in C-peptide levels relative to baseline 2 hours after meals | Week 26
Adverse events (AE) | Week 26
ADA of SHR20004 | Week 26
Nab of SHR20004 | Week 26
The concentration of SHR20004 in plasma at steady state | Week 26

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Chaoyang Hospital Affiliated to Capital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided